CLINICAL TRIAL: NCT06170541
Title: Ultra-High Resolution Computed Tomography (CT) vs. Conventional CT for Detecting Obstructive Coronary Artery Disease (CAD) The CORE-COMPARE Pilot Study
Brief Title: CORE-COMPARE Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00234130
Record Dates: First submitted 2021-03-24; First posted 2023-12-14 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Coronary Heart Disease (CHD)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: blinded, prospective single-center study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- UHR-CT (Ultra-High-Resolution Computed Tomography-Aquilion Precision) (Experimental): Participants in this arm undergo CT scans using the Ultra-High-Resolution CT imaging modality.
  Interventions: Device: Aquilion Precision
- CR-CT (Conventional Resolution Computed Tomography) (Active Comparator): Participants in this arm receive CT scans using the Conventional Resolution CT imaging modality.
  Interventions: Device: Conventional Computed Tomography

INTERVENTIONS:
Device: Aquilion Precision — Ultra-High Resolution CT (UHR CT) capable of resolving anatomy as small as 150 microns, providing CT image quality with resolution typically seen only in cath labs. The UHR detector is newly designed to provide more than twice the resolution when compared with today's CT technology, with an all-new detector as well as tube, gantry and reconstruction technologies.
  Arms: UHR-CT (Ultra-High-Resolution Computed Tomography-Aquilion Precision)
Device: Conventional Computed Tomography — Conventional reconstruction Computed Tomography (CT) represents a pivotal approach in medical imaging.
  Arms: CR-CT (Conventional Resolution Computed Tomography)

SUMMARY:
The utility of Ultra High-Resolution Computed Tomography (UHR-CT) compared to conventional CT in all-comers (i.e., a generally lower-risk population) remains uncertain but is an important area of study in order to justify wider spread implementation and use of this technology, particularly in light of reports of significantly higher radiation exposure with UHR-CT, as well as longer scan times. The availability of technology to reconstruct conventional resolution (CR) simulation images from the raw CT acquisition data acquired on the UHR-CT scanner offers a unique platform to study this question without subjecting individuals to two different scans.

The primary objective of this study is to generate preliminary data in support of the hypothesis that noninvasive UHR-CT is superior to conventional resolution CT for identifying patients with obstructive CHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21-85 years
* Clinical history suggestive of CHD who are referred by their primary cardiologist for further evaluation via Computed tomography angiography (CTA) will be asked to participate.
* Women of child bearing potential must demonstrate a negative pregnancy test within 24 hours of the study CTA.
* Ability to understand and willingness to sign the Informed Consent Form.

Exclusion Criteria:

* Known allergy to iodinated contrast media.
* History of multiple myeloma or previous organ transplantation
* Elevated serum creatinine (> 1.5mg/dl) OR calculated creatinine clearance of < 60 ml/min (using the Cockcroft-Gault formula
* Atrial fibrillation or uncontrolled tachyarrhythmia, or advanced atrioventricular block (second or third degree heart block)
* Evidence of severe symptomatic heart failure (NYHA Class III or IV);
* Known or suspected moderate or severe aortic stenosis
* History of prior percutaneous coronary intervention (PCI) in one or more vessel or history of coronary arterial bypass grafting (CABG)
* Suspected acute coronary syndrome
* Presence of any other history or condition that the investigator feels would be problematic

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2027-04-05 (Estimated)

PRIMARY OUTCOMES:
agreement between the number of patients with >70% stenosis detected by ultra-high-resolution tomography compared to conventional tomography, with catheterization considered as the gold standard. | Up to 24 Months
  The ultra-high-resolution CT images (UHRCT) and the reconstructed conventional CT resolution images (CRCT) will be independently reviewed by two observers (with a 60-day washout period between both images). The stenoses will be classified according to the Society of Cardiovascular Computed Tomography (SCCT) classification system (<25%, 25-49%, 50-69%, 70-99%, and occluded). Patients with stenosis greater than 70% will be flagged.
  The primary outcome will be assessed for patients that underwent a clinically indicated invasive angiography (ICA).
  To compare agreement between UHRCT and CRCT studies while using ICA as the gold-standard, a concordance meta-analysis will be employed. This involves evaluating the agreement measures from each study, standardizing the results, and then comparing the concordance results of the two studies with the third study, considered the gold standard.

SECONDARY OUTCOMES:
Segment-Based Analysis for Obstructive Stenosis: | Up to 24 Months
  Stenosis greater than 70% and 50-69% will be identified and flagged in both imaging modalities (UHRCT and CRCT). The agreement in identifying these specific levels of stenosis will be compared.
Diagnostic Confidence Assessment: | Up to 24 Months
  Confidence level will be classified by the 2 observers for both imaging modalities using the following scale: 1. Very Unsure, 2. Unsure, 3. Moderately Confident, 4. Confident, 5. Highly Confident.
Interobserver Variability Analysis: | Up to 24 Months
  The agreement in the stenosis classification at patient and vessel level will be assessed using Cohen's kappa statistic.
Assessment of vascular and plaque metrics: | Up to 24 Months
  A comparison will be performed between both imaging modalities for the following parameters: vessel volume, lumen volume, wall/lumen ratio, total plaque volume, percentage of calcified component, percentage of non-calcified component.
Pericoronary Adipose Tissue Analysis: | Up to 24 Months
  The perivascular fat attenuation index (FAI) will be calculated for all the three major vessels, right coronary artery (RCA), left circumflex artery (LCX) and left anterior descending (LAD) in both datasets and the results will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Joao Lima, Professor, Principal Investigator — MD
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 12 months after article publication. Data will be made accessible up to 24 months with extensions considered as needed.
Access Criteria: Access provided upon request.